CLINICAL TRIAL: NCT07365007
Title: Feasibility of a Virtually Delivered LASO-3 Diet Intervention for Chemotherapy-Induced Peripheral Neuropathy in Post-Treatment Cancer Survivors
Brief Title: A Virtually Delivered Diet Intervention (LASO-3) for the Improvement of Chemotherapy-Induced Peripheral Neuropathy in Cancer Survivors Post-treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: The Hope Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2025.077; NCI-2025-07988 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HUM00274541 (Other: University of Michigan)
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy; Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Specimen Handling; Early Intervention, Educational; Educational Status; Methods; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (LASO-3 sessions) (Experimental): Patients attend virtual LASO-3 nutrition counseling sessions over 30 minutes QW for 4 weeks followed by LASO-3 nutrition counseling sessions over 15 minutes Q2W for 8 weeks. Patients also undergo blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Interview; Other: Survey Administration
- Arm II (general health education sessions) (Active Comparator): Patients attend eight virtual general health education sessions over 15-30 minutes each over 12 weeks. Patients also undergo blood sample collection throughout the trial. Patients may also receive the intervention materials and up to 4 dietary counseling sessions post-study.
  Interventions: Procedure: Biospecimen Collection; Other: Educational Intervention; Other: Electronic Health Record Review; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Educational Intervention — Attend virtual general health education sessions
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm II (general health education sessions)
Other: Electronic Health Record Review — Ancillary studies
Other: Interview — Ancillary studies
  Arms: Arm I (LASO-3 sessions)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial studies whether a virtually delivered diet intervention focused on lower added sugar, higher fiber, and higher omega 3 fatty acid (LASO-3) can be used to improve chemotherapy-induced peripheral neuropathy (CIPN) in cancer survivors after treatment. Cancer survivors often experience CIPN during and after cancer treatment with neurotoxic chemotherapy. CIPN is characterized by nerve damage from chemotherapy that leads to numbness, tingling, or pain in the hands or feet. However, there are few treatments to manage CIPN. Inflammation contributes to the development of CIPN and dietary patterns that have been demonstrated to improve diet quality and reduce inflammation in cancer survivors may be promising for use as a CIPN management strategy. The LASO-3 diet intervention consists of virtually delivered nutrition education sessions provided by a Registered Dietitian. The sessions focus on three dietary goals, informed by the United States Dietary Guidelines for Americans: 1) lowering added sugar intake to < 10% of daily calories, 2) increasing daily fiber intake to ≥ 20 grams, and 3) increasing intake of moderate-high omega-3 seafood to three or more servings weekly or 3300-3400 mg/day of alpha-linolenic acid (e.g., plant-based sources include canola or flaxseed oil, walnuts, or flaxseed or chia seeds). The Registered Dietitian tailors the sessions to the patient based on information and feedback obtained throughout the sessions. The LASO-3 diet intervention may be an effective way to improve CIPN in cancer survivors after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* At least three months since last receiving neurotoxic chemotherapy
* Self-report moderate (≥ 2/4) numbness and tingling on the Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE™) Numbness and Tingling Severity Item in the last week
* Speak/read English
* Have access to the internet

Exclusion Criteria:

* Pre-existing neuropathy from any cause
* Plan to begin a new prescription of duloxetine (i.e., first-line treatment for CIPN pain) during the study period
* Are enrolled in symptom management trials that may alter CIPN severity
* Current inflammatory disease
* Routine nonsteroidal anti-inflammatory drug (NSAID) or steroid supplementation
* Consuming an average three or more servings of fish per week and/or consuming fish oil capsules containing eicosapentaenoic acid (EPA)+ docosahexaenoic acid (DHA) daily or consuming flax oil capsules daily
* Consuming an average of less than 5 servings of sweets, candy bars, chocolate, doughnuts, cookies, cakes, pie, brownies, ice cream, pastries, or sugar sweetened beverages (e.g., soda or coffee/tea) per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment of all participants (Feasibility) | Up to 2 years
  Feasibility will be established if the following benchmark is met, recruitment of all participants within a two-year period (Demand). The observed recruitment rate will be estimated along with exact 80% confidence intervals (CIs).
Completion of baseline and 12-week patient-reported outcome measures (Feasibility) | At baseline and 12 weeks
  Feasibility will be established if the following benchmark is met, ≥ 60% completion of baseline and 12-week patient-reported outcome measures. The observed retention rate will be estimated along with exact 80% CIs.
Percent of LASO-3 participants who attend at least 5 out of 8 intervention sessions (Feasibility) | Up to 12 weeks
  Feasibility will be established if the following benchmark is met, ≥ 60% of LASO-3 participants attend at least 5 out of 8 intervention sessions (Implementation). The observed retention rate will be estimated along with exact 80% CIs.
Percent of LASO-3 participants who self-report adherence to dietary goals (Feasibility) | Up to 24 weeks
  Feasibility will be established if the following benchmark is met, ≥ 60% of LASO-3 participants self-report adherence to dietary goals via VioScreen food frequency questionnaire and/or monthly adherence checklists (Practicality). The observed adherence rate will be estimated along with exact 80% CIs.

SECONDARY OUTCOMES:
Acceptability and satisfaction with the twelve-week LASO-3 diet intervention | At 12 weeks
  Will determine the LASO-3 diet group participants' perspectives of acceptability and satisfaction with the twelve-week intervention using semi-structured interviews. Semi-structured interviews will be professionally transcribed and analyzed using inductive content analysis. Transcripts will be uploaded to NVivo (QSR International), where Dr. Knoerl and the research team will independently derive codes, collaboratively group them into categories, and identify key themes with representative quotations.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knoerl, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
we will only share de-identified data with others upon reasonable request